CLINICAL TRIAL: NCT06021691
Title: A Cohort Study on the Impact of Gestational Blood Glucose Management and Postnatal Nurturing Environment on Delayed Language Development in Children
Brief Title: Gestational Diabetes Mother-infant Cohort
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gansu Provincial Maternal and Child Health Care Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NCRCCHD-2022-GP-17
Record Dates: First submitted 2023-06-07; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy; Cognitive Impairment; Cohort Study
Keywords: Child cognitive impairment; Intrauterine high-glucose environment; Acquired nurture environment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collection of maternal peripheral blood during pregnancy and umbilical cord blood at delivery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gestational diabetes offspring cohort: The Gestational diabetes(GDM) offspring cohort is to learn about language development assessment in 2-year-old children and causal association with their mother who diagnosed GDM
  Interventions: Behavioral: Acquired nurturing environment
- Healthy maternal offspring cohort: Healthy maternal offspring cohort is to learn about language development assessment in 2-year-old children and causal association with their health mother
  Interventions: Behavioral: Acquired nurturing environment

INTERVENTIONS:
Behavioral: Acquired nurturing environment — Superimposed effects of intrauterine high-sugar environment exposure and postnatal nurturing environment exposure

SUMMARY:
The bi-directional dynamic cohort study is to learn about the effects of prenatal exposure to high blood glucose levels and postnatal nurturing environment factors on delayed language development in children. The study investigated the results of blood glucose screening during pregnancy for the children's mothers, and followed up on the blood glucose management effectiveness of pregnant women with abnormal blood glucose levels before delivery. Participants will be also surveyed the "S-S method for language development assessment, "gsell Scale", and "0-6 year-old family nurturing environment evaluation scale" to evaluate the language development and family nurturing environment.

DETAILED DESCRIPTION:
Glucose management during pregnancy and the postnatal nurturing environment are keys to early detection and early intervention of language delay, which is important to reduce abnormal language development in children. In this study, mothers diagnosed with gestational diabetes mellitus in the department of hospital and offspring were used as participants. The investigators take a follow-up visit to participants' offspring using the S-S method of language development assessment, gsell Infant and Toddler Development Scale, and 0-6 years old family parenting environment evaluation scale. The bi-directional dynamic cohort study is to learn about the effects of prenatal exposure to high blood glucose levels and postnatal nurturing environment factors on delayed language development in children.

ELIGIBILITY:
Inclusion Criteria:

* Children 1.5-2.5 years old with no serious underlying diseases and no hearing impairment.

Exclusion Criteria:

* diagnosed hearing impairment, organic dysarthria, oral disease; (ii) cerebral palsy;
* neurological and hereditary metabolic diseases; (iv) deaf father/mother.

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The pregnant women with abnormal blood glucose levels and the offspring
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
delayed language development in children | 2023.1-2025.11
  "Number of participants diagnosed with GDM," "Number of offspring of participants who participated in the survey of family nurturing environments," and "Composition ratio of offspring with GDM who presented with language delays."

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Wang, Principal Investigator — Gansu Provincial Maternal and Child Health Care Hospital
Locations (1):
- GansuPMCH, Lanzhou, Gansu, China

DOCUMENTS (1):
  • Study Protocol (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT06021691/Prot_000.pdf